CLINICAL TRIAL: NCT06564857
Title: Remifentanil Versus Rocuronium for Optimizing Video Laryngoscopy-assisted Tracheal Intubation in Patients Undergoing General Anaesthesia - a Multicentre Randomised Controlled Trial -The ROCVIDEO Trial
Brief Title: Remifentanil Versus Rocuronium for Optimizing Video Laryngoscopy-assisted Tracheal Intubation
Acronym: ROCVIDEO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ROCVIDEO; 2025-521405-40-01 (EU CTIS Number)
Record Dates: First submitted 2024-06-25; First posted 2024-08-21 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Tracheal Intubation; Video Laryngoscopy; Remifentanil; Rocuronium
MeSH Terms: interventions — Remifentanil; Sodium Chloride; Rocuronium

STUDY DESIGN:
Intervention Model Description: Parallel Assignment, multicenter
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REMI-arm (Experimental): Bolus of remifentanil at anaesthesia induction
  Interventions: Drug: Remifentanil
- ROCU-arm (Active Comparator): Bolus of rocuronium at anaesthesia induction
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Remifentanil — Age < 70 years: Bolus of 4 μg/kg Ideal Body Weight remifentanil at anaesthesia induction; Age >= 70 years: Bolus of 2 μg/kg ideal Body Weight remifentanil at anaesthesia induction
  Other Names: Remifentanil 5 mg diluted in 100 ml saline, which corresponds to Remifentanil 50 micrograms/ml
  Arms: REMI-arm
Drug: Rocuronium — Bolus of 0.6 mg/kg Ideal Body Weight rocuronium at anaesthesia induction
  Other Names: Rocuronium 10 mg/ml
  Arms: ROCU-arm

SUMMARY:
Globally, we are approaching 1 million surgical procedures each day. Tracheal intubation is the mainstay of securing the patient's airway and breathing during general anaesthesia. Approximately 100.000 tracheal intubations are performed annually in Denmark. Airway management remains the primary reason for anaesthesia-related morbidity and mortality. It has been traditionally accepted that best tracheal intubation conditions are obtained by paralysing the patient's muscles, including vocal cords, using a neuromuscular blocking agent (NMBA) such as rocuronium. However, using NBMA may increase the risk of pulmonary complications, intra-operative awareness, in which the patient is paralysed but awake during surgery, anaphylaxis, and re-intubation. In addition, there is a risk of residual neuromuscular blockade postoperatively. In the US, prolonged ventilation and unplanned intubation are the top two most costly perioperative complications. An alternative to NMBA is a large dose of opioids to depress laryngeal reflexes during intubation. The most commonly used non-NMBA modality includes bolus administration of remifentanil. However, remifentanil may cause bradycardia and hypotension. Even short periods of hypotension have been shown to increase the risk of myocardial injury and other serious adverse events such as renal failure, delirium, and even mortality.

Evidence also indicates that intubation conditions using only opioids to facilitate intubation, including remifentanil, are inferior to NMBA. However, these trials are underpowered to assess effects on patient-important outcomes and are mostly at high risk of bias. A recent trial has suggested that remifentanil intubation conditions may not be very different. Almost all existing research comparing NMBA to opioids has focused on intubation conditions for direct laryngoscopy using a conventional Macintosh laryngoscopy blade. In recent years, the implementation and availability of the video laryngoscope have grown exponentially and become universal. The video laryngoscope has vastly improved the ease of tracheal intubation, and the number of failed intubations has decreased by two-thirds in Denmark, where a rapid implementation of the video laryngoscope took place. However, limited evidence exists on whether NMBA improves intubation conditions compared to remifentanil when performing video laryngoscope-assisted tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years
* Undergoing general anaesthesia requiring oro-tracheal intubation
* Absence of indication for rapid sequence induction
* American Society of Anesthesiologists (ASA) physical status score I - III

Exclusion Criteria:

* Known allergies or contraindications to rocuronium (e.g. neuromuscular disease) or remifentanil
* Awake intubation
* Double-lumen endotracheal tube
* Oral, pharyngeal, and laryngeal surgery
* Surgical contraindication for NMBAs (e.g. use of nerve stimulator)
* Patients who are pregnant or breastfeeding
* Patients who do not understand Danish or are unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2648 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with one or more intubation or anaesthesia related adverse events | 0 minutes to 24 hours after administration of drugs for intubation
  Early (< 10 min): Cardiac arrest; anaphylaxis; pulmonary aspiration of gastric content; serious traumatic airway injury; desaturation (SAT < 90%); major hemodynamic instability (MAP < 50, new onset bradycardia < 40 beats/min); or sustained new arrhythmia (causing hemodynamic instability or requiring intervention).
  Late (< 24 h): Death; brain damage including stroke; acute myocardial infarction; ICU admission; re-intubation; respiratory failure (oxygen demand > 5 l/min or requiring interventions aside from oxygen therapy); intraoperative awareness; pneumonia; dental injury; sore throat; or hoarseness.
Proportion of participants with failed first-pass intubation | Tracheal intubation is performed 2 minutes after administration of rocuronium or remifentanil.
  Defined as failed tracheal tube delivery after the first attempt of introduction of the video laryngoscope into the patient's mouth.
  Tracheal tube delivery is defined as failed when the tube is retracted out of the patient's mouth, OR the video laryngoscope has to be retracted out of the patient's mouth, OR there is a shift in intubation equipment OR a change in the person performing the intubation management OR the intubation is abandoned.

SECONDARY OUTCOMES:
Patient satisfaction score | 24 hours after administration of drugs for intubation
  The patient's experience of the treatment using a numeric rating scale (NRS 0 - 10 (0 = very dissatisfied; 10 = very satisfied))
Proportion of participants with one or more serious adverse events 0-7 days | 0 minutes to 7 days after administration of drugs for intubation
  Defined as: respiratory failure, major adverse cardiac (in-hospital all-cause death, acute myocardial infarction (AMI) both acute ST elevation MI and non-ST elevation MI, complete heart block, cardiogenic shock, cardiac arrhythmia and cardiac arrest), pneumonia, acute kidney injury, admission to ICU and cerebrovascular event (ischemic stroke including transient cerebral ischemia).
Lengths of stay at the Post-Anaesthesia Care Unit. | 0-48 hours postoperatively
  Minutes the patient is at the Post-Anaesthesia Care Unit.

OTHER OUTCOMES:
Proportion of participants with failed intubation | 2 to 20 minutes after administration of drugs for intubation
  The intubation is abandoned
Number of intubation attempts | 2 to 20 minutes after administration of drugs for intubation
  The first attempt is defined as an attempt (successful or not) at tracheal tube delivery after the first introduction of the video laryngoscope into the patient's mouth.
  Additionally attempts are defined as: when the tube has to be re-introduced into the patient's mouth, OR the videolaryngoscopy has to be re-introduced into the patient mouth, OR there is a shift in intubation equipment OR a change in the person performing the intubation management
Vocal cords position at first intubation attempt | 2 to 20 minutes after administration of drugs for intubation
  Categorised as closed, intermediate or open
Proportion of participants with need for rescue medication or airway management | 2 to 20 minutes after administration of drugs for intubation
  Rescue medication is defined as: An additional bolus of neuromuscular blocking agents, or bolus of opioid or propofol or other anesthetics according to the discretion of the attending anaesthesiologist in order to solve insufficient airway management conditions.
Proportion of participants with anaesthesia induction related grave desaturation | 0 to 10 minutes after administration of drugs for intubation
  SAT < 80%
Proportion of participants in need of vasoactive or chronotropic substances after induction | 0 to 10 minutes after administration of drugs for intubation
  Defined as any vasoactive substance, e.g. epinephrine, noradrenaline, phenylephrine, ephedrine administrated as a response to severe hypotension or bradycardia after induction.
Individual components of the composite outcomes "Proportion of participants with one or more intubation or anaesthesia related adverse events" and "Proportion of participants with one or more serious adverse events 0-7 days" | 0 minutes to 7 days after administration of drugs for intubation
  As stated in the relevant outcome descriptions

CONTACTS AND LOCATIONS:
Overall Officials: Anders K Nørskov, PhD, Principal Investigator — Department of Anaesthesia, Nordsjællands Hospital - Hillerød, Denmark; Matias Vested, PhD, Principal Investigator — Department of Anaesthesia Centre of Head and Orthopedics Rigshospitalet, University of Copenhagen
Locations (2):
- Denmark (2):
  - Department of Anesthesiology, NOH, Rigshospitalet, Copenhagen
  - Department of Anesthesiology, North Zeeland Hospital, Hillerød

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The protocol is submitted prior to first randomisation. A comprehensive statistical analysis plan, including pre-specified subgroup analysis will be published before the final participant is enrolled.
  Other material will be made available <12 months after trial cessation
Access Criteria: Anonymised data will be made available upon reasonable request.